CLINICAL TRIAL: NCT00174954
Title: A Study to Validate Magnetic Resonance Imaging (MRI) in the Quantitative Assessment of Gouty Tophi.
Brief Title: Magnetic Resonance Imaging in Subjects With Gouty Tophi
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sr. VP, Clinical Science, Takeda Global Research & Development Center, Inc.
Other Study IDs: TMX-01-013; U1111-1113-9856 (Registry Identifier: WHO)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2009-07-16 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Hyperuricemia; Gout
Keywords: Gout; Tophus; MRI
MeSH Terms: conditions — Hyperuricemia; Gout

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: None Retained — None taken or retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Volumes/measurements of tophi determined by serial MRIs
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — Subjects underwent MRI to evaluate tophi.

SUMMARY:
The purpose of this study is to determine the reproducibility of Magnetic Resonance Imaging (MRI) in the quantitative assessment of tophus volume.

DETAILED DESCRIPTION:
This is a multi-center, validation study of MRI in the quantitative assessment of gouty tophi. Subjects with palpable gouty tophi (confirmed by aspiration of the tophus) in select anatomical sites (foot, hand or elbow) will undergo pre- and post contrast MRI on two occasions separated by 5 to 10 days. This study will consist of up to 4 study visits.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with gout and at least one tophi.

Exclusion Criteria:

* Unable to undergo MRI.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with palpable gouty tophi.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2002-03; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Takeda

REFERENCES:
- [Result] Schumacher HR Jr, Becker MA, Edwards NL, Palmer WE, MacDonald PA, Palo W, Joseph-Ridge N. Magnetic resonance imaging in the quantitative assessment of gouty tophi. Int J Clin Pract. 2006 Apr;60(4):408-14. doi: 10.1111/j.1368-5031.2006.00853.x. PMID 16620352
- See also: Uloric Package Insert — http://general.takedapharm.com/content/file.aspx?applicationcode=6C7C39D8-5D09-453B-BF30-696A4AB88E62&fileTypeCode=ULORICPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 6 study centers from 07 March 2002 to 28 January 2003.
Pre-assignment Details: Subjects with palpable gouty tophi in select anatomical sites underwent pre- and post-contrast Magnetic Resonance Imaging (MRI)
Groups:
- Palpable Gouty Tophi Subjects: Volumes/measurements of tophi determined by serial MRI
Period: Overall Study
Arm/Group | Palpable Gouty Tophi Subjects
Started | 32
Completed | 28
Not Completed | 4
Not completed — Adverse Event | 2
Not completed — No tophi found in MRI | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Palpable Gouty Tophi Subjects
Number analyzed (Participants) | 32
Age Continuous [Mean (Standard Deviation); unit: years] | 61.2 (15.5)
Age, Customized [Number; unit: participants]
  18 years to 35 years | 1
  36 years to 50 years | 9
  51 years to 65 years | 7
  66 years to 85 years | 13
  >85 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 30
Race/Ethnicity [Number; unit: participants]
  White | 22
  Black or African American | 9
  Hispanic | 1

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Tophi by MRI - Difference in Volument Between Visits
Description: Two independent readers determined volume of the same tophus by MRI at 2 separate visits scheduled no more than 10 days apart. Difference in volume between Visit 1 and 2 for the same tophus was pooled across readers.
Time Frame: Visit 1 (Day 1) and Visit 2 (Days 6-11)
Population: Analysis was performed on the subjects with MRI tophus volume measurements at both visits from the same reader. Change in tophus size over 10 days was not expected.
Measure: Mean (Standard Deviation); unit: centimeters³ (cm³)
Arm/Group | Palpable Gouty Tophi Subjects
Number analyzed (Participants) | 30
centimeters³ (cm³)
  Mean Difference | -0.05 (0.97)
Statistical Analysis 1: Comparison: Palpable Gouty Tophi Subjects; Test type: Superiority or Other; p = 0.785, paired t-test — The a priori threshold for statistical significance was 0.05

2. Primary Outcome: Measurement of Tophi by MRI - Difference in Volume Between Readers
Description: Two independent readers determined volume of the same tophus by MRI at 2 separate visits scheduled no more than 10 days apart. Difference in Reader 2 volume and Reader 1 volume for the same tophus were pooled across visits.
Time Frame: Visit 1 (Day 1) and Visit 2 (Days 6-11)
Population: Analysis was performed on the subjects with MRI tophus volume measurements from both readers at the same visit.
Measure: Mean (Standard Deviation); unit: cm³
Arm/Group | Palpable Gouty Tophi Subjects
Number analyzed (Participants) | 32
cm³ | 0.89 (2.05)
Statistical Analysis 1: Comparison: Palpable Gouty Tophi Subjects; Test type: Superiority or Other; p = 0.020, paired t-test — The a priori threshold for statistical significance is 0.05

ADVERSE EVENTS:
Arm/Group | Palpable Gouty Tophi Subjects
Serious Adverse Events (participants affected / at risk) | 2/32
Other Adverse Events (participants affected / at risk) | 6/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palpable Gouty Tophi Subjects (N=32)
Rate and Rhythm Disorders not elsewhere classified (NEC) (Cardiac disorders) | 1
Renal Failure and Impairment (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Palpable Gouty Tophi Subjects (N=32)
Gastrointestinal Atonic and Hypomotility Disorders NEC (Gastrointestinal disorders) | 1
Nausea and Vomiting Symptoms (Gastrointestinal disorders) | 1
Febrile Disorders (General disorders) | 1
Muscle Related Signs and Symptoms NEC (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and Connective Tissue Signs and Symptoms NEC (Musculoskeletal and connective tissue disorders) | 1
Nasal Congestion and Inflammations (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.